CLINICAL TRIAL: NCT04946604
Title: Ashtangayoga for IBS Show Positive Preliminary Effects on Symptoms and Well-being in an Uncontrolled Pilot Study
Brief Title: Ashtangayoga for IBS Show Positive Preliminary Effects on Symptoms and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Praktikertjänst AB (Ltd) (Other)
Responsible Party: Principal Investigator, Perjohan Lindfors, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 751-17
Record Dates: First submitted 2021-06-08; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Each participant is given the intervention, and they are measured at pre, post and 6 month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ashtangayoga (Other): Participants attanded eight yoga sessions, one hour long.
  Interventions: Behavioral: Ashtangayoga

INTERVENTIONS:
Behavioral: Ashtangayoga — This is an active and intense type of yoga, focused on physical activity and breath control

SUMMARY:
The study aims to test the effect of Ashtanga yoga on well-being in patients with irritable bowel syndrome (IBS). The intervention comprises group sessions on the Ashtanga school of yoga. Participants are recruited from primary care and measurements on well-being and IBS symptoms are conducted at pre-treatment, post-treatment and 6-month follow-up.

DETAILED DESCRIPTION:
The intervention comprises participants with IBS to undergo Ashtanga yoga sessions in a group led by an authorized yoga teacher for a total period of 10 weeks. The first 4 weeks consisted of 1 session/week and the following 6 weeks consisted of 1 session/2 weeks. All movements and exercises are performed based on the individual's personal capacity in order to avoid distinct discomfort or pain. Patients testing positive for IBS will be recruited for the study from primary care. Measurements of IBS symptoms, visceral sensitivity, extraintestinal symptoms and quality of life will be assessed at pre-treatment, post-treatment and 6-month follow-up. Specific statistical methods will be performed to assess changes from pre- to post-treatments and changes from post-treatment to 6-month-follow-up. Effects sizes for within group changes will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosis

Exclusion Criteria:

* Prior yoga practise, unable to speak Swedish, other serious illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) | Change from pre-treatment (baseline) to post-treatment (week 10), change from post-treatment (week 10) to follow-up (week 22)
  Irritable Bowel Syndrome Severity Scoring System (IBS-SSS; [17] is a scale that measure the global severity of IBS-symptoms. It includes five items; pain severity, pain frequency, bowel bloating, bowel habit dissatisfaction and life interference that are scored on a visual analogue scale (VAS) 0-100 mm. The total score ranges from 0-500 with higher scores indicating more severe symptoms.
Change in Gastrointestinal Symptom Rating Scale - IBS version (GSRS-IBS) | Change from pre-treatment (baseline) to post-treatment (week 10), change from post-treatment (week 10) to follow-up (week 22)
  Gastrointestinal Symptom Rating Scale - IBS version (GSRS-IBS; [18] measures the severity of IBS-symptoms experienced over the past week. The scale consists of 13 items measuring five symptom domains of IBS: satiety, pain, diarrhea, constipation and bloating. The symptoms are rated on a scale ranging from 1 (= no discomfort) to 7 (= very severe discomfort) with a total score from 13-91. Higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
IBS Quality of Life (IBSQOL) | Pre (0 weeks), post (after 10 weeks), follow-up (after 22 weeks)
  IBS Quality of Life (IBSQOL; [19] is a disease-specific health-related quality of life scale (HRQOL). The instrument consists of 34 items that measure nine domains of quality of life: emotional functioning, mental health, physical functioning, sleep, diet, energy, social role, physical role and sexual relations. Each item is rated on a scale from 1 to 5 or 1 to 6, the raw scores is then transformed into a scale of 0-100 with higher scores indicating a better IBS-specific quality of life.
Visceral Sensitivity Index (VSI) | Pre (0 weeks), post (after 10 weeks), follow-up (after 22 weeks)
  Visceral Sensitivity Index (VSI; [20] measures gastrointestinal symptom-specific anxiety. The scale consists of 15 items rated on a scale from 0 (=strongly agree) to 5 (=strongly disagree). The total score ranges from 0-75 with higher scores suggesting higher GI-related anxiety
Hospital Anxiety and Depression Scale (HADS) | Pre (0 weeks), post (after 10 weeks), follow-up (after 22 weeks)
  Hospital Anxiety and Depression Scale (HADS; [21] measures the severity of anxiety and depression in non-psychiatric patients. It consists of 14 items, seven related to anxiety and seven to depression. Each item is scored from 0-3 which gives a total range of 0-21 points. Higher scores indicate more severe symptoms.
The Patient Health Questionnaire 12 (PHQ-12) | Pre (0 weeks), post (after 10 weeks), follow-up (after 22 weeks)
  The Patient Health Questionnaire 12 (PHQ-12; [22] is a modification of PHQ-15 which measures the experience of 15 different somatic symptoms. Three of the 15 items are GI-related and are therefore excluded from the PHQ-12 in order to be able to exclusively measure extraintestinal somatic symptoms. The symptoms measured are back pain, chest pain, dizziness, fainting spells, feeling the heart pound or race, headaches, pain in arms or legs, pain during sexual intercourse, shortness of breath, tiredness, trouble sleeping and problems with the period. The questionnaire consists of 12 items rated on a scale from 0 (=not bothered at all) to 2 (=bothered a lot). The total score ranges from 0-24, higher scores indicate greater extraintestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Perhjohan Lindfors, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Centre for psychatry research, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No